CLINICAL TRIAL: NCT06954805
Title: Defining the Role of ctDNA Monitoring in a Risk Stratified Clinical Trial for Posttransplant Lymphoproliferative Disorder (PTLD)
Brief Title: Defining ctDNA Metrics in Posttransplant Lymphoproliferative Disorder (PTLD)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jennifer Amengual (Other)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor-Investigator, Jennifer Amengual, Associate Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAV2404
Record Dates: First submitted 2025-04-24; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Lymphoma; Lymphoma, B-Cell
Keywords: posttransplant; lymphoproliferative disorder
MeSH Terms: conditions — Lymphoma; Lymphoma, B-Cell; Lymphoproliferative Disorders | interventions — Rituximab; Etoposide; etoposide phosphate; Prednisone; Vincristine; Cyclophosphamide; Doxorubicin; Biological Assay

STUDY DESIGN:
Intervention Model Description: All participants will receive induction therapy consisting of 4 weekly cycles of rituximab. Following completion of induction therapy, participants will be risk stratified into one of two different consolidative treatment regimens based on whether they qualify as either low-risk or high-risk. Risk stratification will be made based on both radiographic response to induction therapy as well as the underlying biologic features of their PTLD.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm A (Low-risk) (Experimental): Following completion of induction therapy, participants will be assigned to Arm A if they meet the following criteria:
  1. Complete response to rituximab induction
     OR
  2. Partial response to rituximab induction without any additional high-risk features.
  Low-risk participants will receive IV rituximab 375 mg/m2 every 21 days for 4 cycles.
  Interventions: Drug: Rituximab; Device: CAPP-seq
- Arm B (High-risk) (Experimental): Following completion of induction therapy, participants will be assigned to Arm B if they meet the following criteria:
  1. Stable disease
  2. Progressive disease
     OR
  3. Partial response to rituximab induction with any of the following:
     * Residual bulky disease, defined as any single lesion measuring ≥ 7 cm or any 3 lesions each measuring ≥ 3 cm
     * High risk cytogenetic features including a complex karyotype (defined as ≥3 abnormalities on conventional karyotype), FISH positive for MYC rearrangement, double hit lymphoma (defined as MYC rearranged with BCL2 or BCL6), or p53 derangements
     * Plasmablastoid histology
  High-risk participants will receive R-EPOCH every 21 days for 4 cycles:
  * Rituximab 375 mg/m2 IV Day 1
  * Etoposide 50 mg/m2 IV Day 1, 2, 3, 4
  * Prednisone 60 mg/m2 PO Day 1, 2, 3, 4, 5
  * Vincristine 0.4 mg/m2 IV Day 1, 2, 3, 4
  * Cyclophosphamide 375 mg/m2 IV Day 5
  * Doxorubicin 10 mg/m2 IV Day 1, 2, 3, 4
  Interventions: Drug: Rituximab; Drug: Etoposide; Drug: Prednisone; Drug: Vincristine; Drug: Cyclophosphamide; Drug: Doxorubicin; Device: CAPP-seq

INTERVENTIONS:
Drug: Rituximab — Rituximab is a genetically engineered chimeric murine/human monoclonal IgG1 kappa antibody directed against the CD20 antigen. The Fab domain of rituximab binds to the CD20 antigen on B lymphocytes, and the Fc domain recruits immune effector functions to mediate B cell lysis. 375 mg/m2 Rituximab will be administered to participants by IV.
Drug: Etoposide — Etoposide is a topoisomerase II inhibitor and appears to cause DNA strand breaks. It has been shown to delay transit of cells through S phase and arrest cells in late S or early G2 phase. 50 mg/m2 Etoposide will be administered to participants by IV.
  Other Names: Etopophos
  Arms: Arm B (High-risk)
Drug: Prednisone — Prednisone can prevent or suppress inflammation and immune responses. Prednisone's action may include the inhibition of leukocyte infiltration at the site of inflammation, interference in the function of mediators of inflammatory response, and suppression of humoral immune responses. 60 mg/m2 Prednisone will be administered to participants by PO.
  Arms: Arm B (High-risk)
Drug: Vincristine — Vincristine is a vinca alkaloid. The mechanism of action of vincristine is thought to be due to inhibition of microtubule formation in the mitotic spindle. This leads to arrest of dividing cells during the metaphase stage. 0.4 mg/m2 Vincristine will be administered to participants by IV.
  Other Names: Oncovin
  Arms: Arm B (High-risk)
Drug: Cyclophosphamide — The mechanism of action is thought to involve cross-linking of tumor cell DNA. Cyclophosphamide is biotransformed principally in the liver to active alkylating metabolites which are thought to cross-link to tumor cell DNA. These metabolites interfere with the growth of rapidly proliferating susceptible malignant cells. 375 mg/m2 Cyclophosphamide will be administered to participants by IV.
  Other Names: Cytoxan
  Arms: Arm B (High-risk)
Drug: Doxorubicin — Doxorubicin is an anthracycline, topoisomerase II inhibitor. It is isolated from cultures of Streptomyces peucetius var. caesius. The cytotoxic effect of doxorubicin is related to nucleotide base intercalation and cell membrane lipid binding activities. It blocks nucleotide replication and the action of DNA and RNA polymerases. The interaction between doxorubicin and topoisomerase II to form DNA-cleavable complexes appears to be an important mechanism of its cytocidal activity. 10 mg/m2 Doxorubicin will be administered to participants by IV.
  Other Names: Adriamycin
  Arms: Arm B (High-risk)
Device: CAPP-seq — Next generation sequencing (NGS) tool used to detect tiny amounts of cancer DNA in the blood, allowing for early diagnosis and monitoring of cancer in a non-invasive way.
  Other Names: cancer personalized profiling by deep sequencing; cell free DNA (cfDNA) assay

SUMMARY:
The purpose of this study is to find out if there is a benefit to giving rituximab with etoposide, prednisone, vincristine, cyclophosphamide and doxorubicin (R-EPOCH) in participants who have high-risk B-cell PTLD in their 2nd phase of treatment (consolidation) while those with low-risk disease will be spared of chemotherapy and treated with rituximab consolidation alone.

This study is also being done to find out about the usefulness of circulating tumor DNA (ctDNA), a novel blood test which, has been shown to help guide treatment decisions in other types of lymphoma. The goal is to answer the question if ctDNA is a viable and informative tool in treating PTLD with the hope that in the future it may be used to individualize study treatment for participants with PTLD in a way that limits study treatment toxicity without losing the effectiveness of the treatment plan.

DETAILED DESCRIPTION:
This is a multi-center, phase 2, open-label clinical trial to evaluate the efficacy of dose modified R-EPOCH in high-risk, treatment naïve CD20+ posttransplant lymphoproliferative disorder (PTLD) patients. The purpose of this study is to define the benefit of rituximab with etoposide, prednisone, vincristine, cyclophosphamide and doxorubicin (R-EPOCH) in patients who have high-risk B cell PTLD while those with low-risk disease will be spared of chemotherapy and treated with rituximab alone. Concurrently this study also seeks to evaluate the usefulness of circulating tumor DNA (ctDNA), a novel blood test which has been shown to improve a physician's ability to prognosticate and guide treatment decisions in other types of lymphoma. The goal is to demonstrate that ctDNA is a viable and informative tool in treating PTLD with the hope that in the future it may be used to individualize treatment for patients with PTLD in a way that limits treatment toxicity without losing the effectiveness of the treatment plan.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed CD20+ PTLD including the below subtypes:

  * Polymorphic
  * Monomorphic
* Age ≥ 15.
* Participants must have measurable disease, defined as lymph node ≥ 1.5 cm in greatest diameter per Lugano Classification
* Patients must have a PET-CT scan (preferred; alternatively CT chest, abdomen and pelvis with IV contrast) performed within 28 days prior to the start of the study.
* All participants must be screened for chronic hepatitis B virus (HBV) within 28 days prior to registration. Participants with known HBV infection (positive serology) must also have a HBV viral load performed within 28 days prior to registration, and participants must have an undetectable HBV viral load on suppressive therapy within 28 days prior to start of treatment. Participants found to be HBV carriers during screening are eligible and must receive standard of care prophylaxis. Participants with active Hepatitis B (HBV viral load > 500 IU/mL) within 28 days prior to registration are not eligible.
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. Participants with an active HCV infection who are currently on treatment must have an undetectable HCV viral load within 28 days prior to registration.
* Participants with known human immunodeficiency virus (HIV)-infection are eligible providing they are on effective anti-retroviral therapy and have undetectable viral load at their most recent viral load test (must be within 26 weeks prior to registration). Participants with known HIV must have a CD4 count checked within 28 days prior to registration, but may proceed with therapy regardless of CD4 count.
* Organ function as assessed by laboratory testing is in appropriate range for receipt of rituximab and R-EPOCH per individual treating physician discretion.
* Cardiac function testing is in appropriate range for receipt of rituximab and R-EPOCH per individual treating physician discretion.
* Eastern Cooperate Oncology Group (ECOG) performance status is in appropriate range for receipt of rituximab and R-EPOCH per individual treating physician discretion.
* Ability to understand and the willingness to sign a written informed consent document. In cases of partial impairment, impairment that fluctuates over time, or complete impairment due to dementia, stroke, traumatic brain injury, developmental disorders (including mentally disabled persons), serious mental illness, and delirium, a subject may be enrolled if the subject's legally authorized representative consents on the subject's behalf.
* Due to the potential teratogenic effects of chemotherapy, women of childbearing age must have a documented negative serum β-hCG measured within 2 weeks of starting treatment.
* Both women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence).
* Women must agree to not breastfeed during the entirety of the study period.
* Participants must not have had chemotherapy for other indications within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study and must have recovered from adverse events due to agents administered more than 4 weeks earlier.
* Participants must not have received more than a cumulative of dose 250 mg/m 2 of prior doxorubicin (or equivalent dose of another anthracycline, such as epirubicin) therapy (at any time prior to registration).
* Intrathecal chemotherapy administered for CNS prophylaxis is allowed in addition to protocol therapy per institution practice.

Exclusion Criteria:

* Patients who have received systemic chemotherapy for PTLD.
* Patients who have known lymphomatous involvement of the central nervous system (CNS).

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2027-04-14 (Estimated); Study Completion 2028-04-14 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Complete Response (CR) rate of 60% or higher | Up to 3 years
  to determine the rate of early molecular response to induction rituximab as well as correlate the experience of undetectable measurable residual disease at mid-consolidation and end of treatment

SECONDARY OUTCOMES:
Circulating tumor DNA (ctDNA) rate | Up to 3 years
  to determine the rate of early molecular response to induction rituximab
Event Free Survival rate | Up to 3 years
  EFS is defined as the duration of time from start of treatment to the time of any treatment failure including disease progression, death, and treatment discontinuation for any reason (e.g., adverse effects or withdrawal).
Duration of Overall Response (OR) | Up to 3 years
  Duration of overall response: The duration of overall response is measured from the time measurement criteria are met for Complete Response (CR) or Partial Response (PR) (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
Duration of stable disease | Up to 3 years
  Stable disease is measured from the start of the treatment until the criteria for progression are met, taking as reference the smallest measurements recorded since the treatment started, including the baseline measurements.
Progression-Free Survival (PFS) rate | Up to 3 years
  PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
Early Molecular Response (EMR) rate | Up to 3 years
  EMR is defined as at least a 2-log fold reduction in circulating tumor DNA (ctDNA) levels between the start and completion of induction therapy.
Measurable Residual Disease (MRD) rate | 8 weeks
  MRD refers to the quantity of ctDNA that can be detected at any given time point following the start of treatment. Undetectable MRD (uMRD) will refer to quantities of ctDNA that fall below the threshold of detection for the CAPP-Seq assay. MRD will be determined by ctDNA assay at both mid-consolidation (between cycles 6 and 7) and EOT (within 8 weeks of C8D1).

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Amengual, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Stanford Medical Center, Stanford, California
  - Columbia University Irving Medical Center, New York, New York